CLINICAL TRIAL: NCT00871377
Title: Pilot Randomized Double Blind Crossover Study Of Fish Oil [Eicosapentaenoic Acid (EPA) And Docosahexaenoic Acid (DHA)] For Intractable Partial Seizures
Brief Title: Double Blind, Crossover Study of Fish Oil [EPA and DHA] for Intractable Partial Seizures
Acronym: FOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, DeGiorgio, Chris, Assistant Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R21AT003420-01A2 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Epilepsy
Keywords: epilepsy; cardiac risk factors; memory; cognition; n-3 fatty acids; fish oil; EPA; DHA; seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Corn Oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Corn Oil Placebo (n-6 fatty acids)
  Interventions: Drug: Placebo
- High Dose Fish Oil (Experimental): 2160 mg of EPA + DHA
  Interventions: Drug: High Dose Fish Oil
- Low Dose Fish Oil (Experimental): 1060 mg of EPA + DHA
  Interventions: Drug: Low Dose Fish Oil

INTERVENTIONS:
Drug: Placebo — corn oil (n-6 fatty acids)
  Other Names: Corn Oil
  Arms: Placebo
Drug: High Dose Fish Oil — n-3 fatty acids, 1060 mg EPA + DHA
  Arms: High Dose Fish Oil
Drug: Low Dose Fish Oil — n-3 fatty acids, 2160 mg EPA + DHA
  Arms: Low Dose Fish Oil

SUMMARY:
The purpose of this study is to determine if Omega-3 fatty acids reduce seizures and modify cardiac risk factors in people with epilepsy.

DETAILED DESCRIPTION:
Epilepsy is a common and disabling condition, characterized by recurrent seizures. Sudden unexpected death (SUDEP) is a major cause of mortality in people with epilepsy. SUDEP accounts for up to 20% of all cause mortality, and is most common in younger people, especially in their 20's to 40's year olds. In those with drug resistant epilepsy, SUDEP is five times more common than in well-controlled epilepsy. Likely causes of death include cardiac arrhythmias due to impaired autonomic regulation and reduced heart rate variability. Similarly, patients with recent myocardial infarction and congestive heart failure are at higher risk for sudden death, and manifest markedly reduced heart rate variability. Clinical studies of heart disease indicate that n-3 fatty acids, prevent cardiac arrhythmias, reduce mortality after myocardial infarction, and reduce the risk of sudden cardiac death. The mechanism by which EPA and DHA exert their anti-arrhythmia effect is due to inactivation of high frequency sodium and L-type calcium channels in the heart. In addition, n-3 fatty acids improve HRV in cardiac patients, and this reduction in HRV is postulated to be a marker of the anti-arrhythmic effect of n-3 fatty acids. Preliminary data from our group indicates that n-3 fatty acids improve HRV in people with epilepsy, especially those with low HRV (SDNN < 50). The commonality between n-3 fatty acids and improvement in HRV in patients with heart disease and epilepsy serves as a basis for our hypothesis that n-3 fatty acids may reduce the risk of SUDEP in epilepsy. The purpose of this proposal is to determine if n-3 fatty acids reduce seizures and modify cardiac risk in people with epilepsy who are at risk of SUDEP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 - 70
* History of intractable localization related/partial onset seizures and generalized tonic/clonic or tonic seizures defined according to International League Against Epilepsy (ILAE) classification as:
* A history compatible with localization related partial epilepsy
* A history of generalized tonic clonic or tonic seizures with loss of consciousness
* Three or more simple partial, complex partial or tonic-clonic seizures per month
* An EEG and/or an MRI consistent with a localization related epilepsy
* Evidence of at least three seizures per month for at least two months prior to the study
* Exposure to at least one antiepileptic drug at adequate dose

Exclusion Criteria:

* Significant or progressive medical, cardiac, or other illness
* Allergy to fish products or fish oil
* History of a coagulation disorder
* History of non-epileptic seizures
* Consumption of Fish Oil at any time 30 days or less prior to enrollment
* Any change in antiepileptic drugs for 30 days or less prior to enrollment
* Treatment with Warfarin for 30 days or less prior to enrollment
* Previous poor compliance with therapy
* Drug or alcohol abuse
* Uncountable seizures as a result of seizure clustering, or inadequate supervision if the patient cannot count their own seizures.
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M DeGiorgio, MD, Principal Investigator — David Geffen - UCLA School of Medicine
Locations (1):
- UCLA General Clinical Research Center, Los Angeles, California, United States

REFERENCES:
- [Background] DeGiorgio CM, Miller P, Meymandi S, Gornbein JA. n-3 fatty acids (fish oil) for epilepsy, cardiac risk factors, and risk of SUDEP: clues from a pilot, double-blind, exploratory study. Epilepsy Behav. 2008 Nov;13(4):681-4. doi: 10.1016/j.yebeh.2008.08.001. Epub 2008 Sep 7. PMID 18721899
- [Background] DeGiorgio CM, Miller P. n-3 fatty acids (eicosapentanoic and docosahexanoic acids) in epilepsy and for the prevention of sudden unexpected death in epilepsy. Epilepsy Behav. 2008 Nov;13(4):712-3. doi: 10.1016/j.yebeh.2008.06.017. Epub 2008 Aug 9. No abstract available. PMID 18634902
- [Result] DeGiorgio CM, Miller P, Meymandi S, Chin A, Epps J, Gordon S, Gornbein J, Harper RM. RMSSD, a measure of vagus-mediated heart rate variability, is associated with risk factors for SUDEP: the SUDEP-7 Inventory. Epilepsy Behav. 2010 Sep;19(1):78-81. doi: 10.1016/j.yebeh.2010.06.011. Epub 2010 Jul 27. PMID 20667792
- [Derived] Novak JL, Miller PR, Markovic D, Meymandi SK, DeGiorgio CM. Risk Assessment for Sudden Death in Epilepsy: The SUDEP-7 Inventory. Front Neurol. 2015 Dec 9;6:252. doi: 10.3389/fneur.2015.00252. eCollection 2015. PMID 26696953
- [Derived] DeGiorgio CM, Miller PR, Harper R, Gornbein J, Schrader L, Soss J, Meymandi S. Fish oil (n-3 fatty acids) in drug resistant epilepsy: a randomised placebo-controlled crossover study. J Neurol Neurosurg Psychiatry. 2015 Jan;86(1):65-70. doi: 10.1136/jnnp-2014-307749. Epub 2014 Sep 8. PMID 25201887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the local epilepsy society, and from flyers posted in the epilepsy clinic at UCLA, and from referrals within the UCLA Department of Neurology
Groups:
- P L H: Placebo, then Low Dose, then High Dose
- P H L: Placebo, then High Dose, then Low Dose
- L H P: Low Dose, then High Dose, then Placebo
- L P H: Low Dose, then Placebo, then High Dose
- H L P: High Dose, then Low Dose, then Placebo
- H P L: High Dose, then Placebo, then Low Dose
Period: First Intervention (10 Weeks)
Arm/Group | P L H | P H L | L H P | L P H | H L P | H P L
Started | 3 | 4 | 4 | 4 | 4 | 5
Completed | 3 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout (6 Weeks)
Arm/Group | P L H | P H L | L H P | L P H | H L P | H P L
Started | 3 | 4 | 3 | 4 | 4 | 4
Completed | 2 | 4 | 3 | 4 | 4 | 4
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (10 Weeks)
Arm/Group | P L H | P H L | L H P | L P H | H L P | H P L
Started | 2 | 4 | 3 | 4 | 4 | 4
Completed | 2 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (6 Weeks)
Arm/Group | P L H | P H L | L H P | L P H | H L P | H P L
Started | 2 | 4 | 3 | 4 | 4 | 4
Completed | 2 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Period: Third Intervention (10 Weeks)
Arm/Group | P L H | P H L | L H P | L P H | H L P | H P L
Started | 2 | 4 | 3 | 4 | 4 | 3
Completed | 2 | 4 | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 Female, 8 Male
Groups:
- Baseline: The study began on Visit 1 when baseline data was collected and Intervention 1 was initiated.
Arm/Group | Baseline
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.04 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency
Description: Seizure frequency (seizures per day or seizures per month)
Time Frame: Study completion (42 weeks)
Measure: Mean (Standard Error); unit: Seizures per Day
Groups:
- Placebo: Corn Oil - 6 capsules per day
- Fish Oil Low Dose: Fish Oil - 3 capsules per day Corn Oil - 3 capsules per day EPA+DHA = 1080 mg/day
- Fish OIl High Dose: Fish Oil - 6 capsules per day EPA+DHA = 2160 mg/day
Arm/Group | Placebo | Fish Oil Low Dose | Fish OIl High Dose
Number analyzed (Participants) | 22 | 20 | 20
Seizures per Day | 0.655 (0.153) | 0.435 (0.097) | 0.631 (0.163)

ADVERSE EVENTS:
Groups:
- High Dose: High Dose Fish Oil Intervention
- Low Dose: Low Dose Fish Oil Intervention
- Placebo: Corn Oil Placebo
Arm/Group | High Dose | Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=20) | Low Dose (N=20) | Placebo (N=22)
Sudden Death in Epilepsy (Cardiac disorders) | 1 (1) | 0 | 0 — 32 year old subject died after a seizure. Found supine on floor next to bed after likely seizure. Autopsy confirmed SUDEP, unrelated to participation in study or study supplement (Fish Oil). Reported to IRB and NIH immediately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No